CLINICAL TRIAL: NCT01536275
Title: Impact of Early Parenteral Nutrition Completing Enteral Nutrition in Paediatric Critically Ill Patients
Brief Title: Early Versus Late Parenteral Nutrition in the Pediatric Intensive Care Unit
Acronym: PEPaNIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Sophia Kindergeneeskunde (Other); Stollery Children's Hospital (Other)
Responsible Party: Principal Investigator, Greet Van den Berghe, Head of Dept Intensive Care Medicine, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEPaNIC; 2012-000811-10 (EudraCT Number); ML8052 (Other: IRB KU Leuven); NL38772.000.12 (Other: IRB CCMO Netherlands); IWT-TBM 110685 (Other Grant/Funding Number: Agency for Innovation by Science & Technology)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Critical Illness; Children
Keywords: critical illness; children; nutrition; metabolism
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early parenteral nutrition (No Intervention): Parenteral nutrition supplements insufficient enteral nutrition from admission to ICU according to the current standard of care per center
- Late parenteral nutrition (Experimental): Parenteral nutrition will be withheld during the first 7 days of ICU stay
  Interventions: Other: Late parenteral nutrition

INTERVENTIONS:
Other: Late parenteral nutrition — Withholding parenteral nutrition during the first 7 days of ICU stay
  Other Names: Late PN
  Arms: Late parenteral nutrition

SUMMARY:
In the PEPaNIC trial it is investigated whether withholding parenteral nutrition during the first week in critically ill children is beneficial, compared to the current standard of the early start of parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the PICU with a STRONGkids score of 2 points or more upon ICU admission

Exclusion Criteria:

* Age of 17 years or older
* Patients with a DNR code at the time of ICU admission.
* Patients expected to die within 12 hours (=moribund patients).
* Patient readmitted to ICU after randomization to the PEPaNIC trial, more than 48 hours after the initial discharge
* Patients transferred from another paediatric intensive care after a stay of more than 7 days
* Patients suffering from ketoacidotic or hyperosmolar coma on admission.
* Patients suffering from Short Bowel Syndrome on home PN or other conditions that require home PN
* Patients suspicious or established inborn metabolic diseases requiring specific diet
* STRONGkids score lower than 2 on ICU admission.
* Premature Newborns ( 37 weeks gestational age upon admission in the PICU)
* Prior inclusion in another randomized controlled outcome study

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1440 (Actual)
Dates: Start 2012-06; Primary Completion 2016-03 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of new infection during ICU stay | during ICU stay and up to 90 days post-randomization
Duration of ICU dependency (crude stay days and time to alive discharge from ICU) | during ICU stay and up to 90 days post-randomization

SECONDARY OUTCOMES:
Mortality | during ICU stay, hospital stay and up to 90 days post-randomization
Time to alive discharge from hospital | during hospital stay and up to 90 days post-randomization
Incidence of hypoglycaemia during ICU stay | during the intervention window up to day 8 post-randomization
Time to final weaning from mechanical respiratory support | during ICU stay and up to 90 days post-randomization
Incidence of liver dysfunction during ICU stay | during ICU stay and up 90 days post-randomization
Need for haemodynamic support during ICU stay | during ICU stay and up 90 days post-randomization
Incidence of new kidney injury during ICU stay | during ICU stay and up 90 days post-randomization
Duration of antibiotics treatment during ICU stay | during ICU stay and up to 90 days post-randomization
Number of readmissions to the ICU | up to 90 days post-randomization
Amount of calories delivered during the ICU stay and in subset markers of feeding intolerance | during the intervention window of 8 days and up to 90 days post-randomization
Markers of inflammation such as C-reactive protein concentrations during ICU stay | during ICU stay and up to 90 days post-randomization
Structural and or functional differences in muscle tissue during ICU stay | during ICU stay and up to 90 days post-randomization
biochemical, metabolic, endocrine, immunological, inflammatory and (epi)genetic markers on blood samples | up to 4 years post-randomization
  with healthy matched control group
functional and neurocognitive development | up to 4 years post-randomization
  with healthy matched control group
health economy analysis | during index hospitalization
  total health care costs during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Greet Van den Berghe, MD PhD, Principal Investigator — KU Leuven
Locations (3):
- Dept Intensive Care Medicine, Leuven, Belgium
- Stollery Children's Hospital, Edmonton, Alberta, Canada
- Erasmus MC Sophia Kinderziekenhuis, Rotterdam, Netherlands

REFERENCES:
- [Background] Casaer MP, Mesotten D, Hermans G, Wouters PJ, Schetz M, Meyfroidt G, Van Cromphaut S, Ingels C, Meersseman P, Muller J, Vlasselaers D, Debaveye Y, Desmet L, Dubois J, Van Assche A, Vanderheyden S, Wilmer A, Van den Berghe G. Early versus late parenteral nutrition in critically ill adults. N Engl J Med. 2011 Aug 11;365(6):506-17. doi: 10.1056/NEJMoa1102662. Epub 2011 Jun 29. PMID 21714640
- [Background] Vlasselaers D, Milants I, Desmet L, Wouters PJ, Vanhorebeek I, van den Heuvel I, Mesotten D, Casaer MP, Meyfroidt G, Ingels C, Muller J, Van Cromphaut S, Schetz M, Van den Berghe G. Intensive insulin therapy for patients in paediatric intensive care: a prospective, randomised controlled study. Lancet. 2009 Feb 14;373(9663):547-56. doi: 10.1016/S0140-6736(09)60044-1. Epub 2009 Jan 26. PMID 19176240
- [Derived] Nakano FK, Dulfer K, Vanhorebeek I, Wouters PJ, Verbruggen SC, Joosten KF, Guiza Grandas F, Vens C, Van den Berghe G. Predicting adverse long-term neurocognitive outcomes after pediatric intensive care unit admission. Comput Methods Programs Biomed. 2024 Jun;250:108166. doi: 10.1016/j.cmpb.2024.108166. Epub 2024 Apr 10. PMID 38614026
- [Derived] Veldscholte K, Hulst JM, Eveleens RD, de Jonge RCJ, de Koning BAE, van den Berg SAA, van der Wal R, Ruijter GJG, Rizopoulos D, Vanhorebeek I, Gunst J, Casaer M, Van den Berghe G, Joosten KFM, Verbruggen SCAT. Gastrointestinal Biomarkers and Their Association with Feeding in the First Five Days of Pediatric Critical Illness. J Pediatr Gastroenterol Nutr. 2023 Dec 1;77(6):811-818. doi: 10.1097/MPG.0000000000003950. Epub 2023 Sep 20. PMID 37728917
- [Derived] Verlinden I, Coppens G, Vanhorebeek I, Guiza F, Derese I, Wouters PJ, Joosten KF, Verbruggen SC, Van den Berghe G. Long-term impact of paediatric critical illness on the difference between epigenetic and chronological age in relation to physical growth. Clin Epigenetics. 2023 Jan 14;15(1):8. doi: 10.1186/s13148-023-01424-w. PMID 36639798
- [Derived] Coppens G, Vanhorebeek I, Verlinden I, Derese I, Wouters PJ, Joosten KF, Verbruggen SC, Guiza F, Van den Berghe G. Assessment of aberrant DNA methylation two years after paediatric critical illness: a pre-planned secondary analysis of the international PEPaNIC trial. Epigenetics. 2023 Dec;18(1):2146966. doi: 10.1080/15592294.2022.2146966. Epub 2022 Nov 16. PMID 36384393
- [Derived] Vanhorebeek I, Jacobs A, Mebis L, Dulfer K, Eveleens R, Van Cleemput H, Wouters PJ, Verlinden I, Joosten K, Verbruggen S, Van den Berghe G. Impact of critical illness and withholding of early parenteral nutrition in the pediatric intensive care unit on long-term physical performance of children: a 4-year follow-up of the PEPaNIC randomized controlled trial. Crit Care. 2022 May 12;26(1):133. doi: 10.1186/s13054-022-04010-3. PMID 35549984
- [Derived] Verlinden I, Guiza F, Dulfer K, Van Cleemput H, Wouters PJ, Guerra GG, Joosten KF, Verbruggen SC, Vanhorebeek I, Van den Berghe G. Physical, Emotional/Behavioral, and Neurocognitive Developmental Outcomes From 2 to 4 Years After PICU Admission: A Secondary Analysis of the Early Versus Late Parenteral Nutrition Randomized Controlled Trial Cohort. Pediatr Crit Care Med. 2022 Aug 1;23(8):580-592. doi: 10.1097/PCC.0000000000002971. Epub 2022 May 9. PMID 35522534
- [Derived] Jacobs A, Guiza F, Verlinden I, Dulfer K, Garcia Guerra G, Joosten K, Verbruggen SC, Vanhorebeek I, Van den Berghe G. Differential DNA methylation by early versus late parenteral nutrition in the PICU: a biological basis for its impact on emotional and behavioral problems documented 4 years later. Clin Epigenetics. 2021 Jul 27;13(1):146. doi: 10.1186/s13148-021-01124-3. PMID 34315515
- [Derived] Verlinden I, Dulfer K, Vanhorebeek I, Guiza F, Hordijk JA, Wouters PJ, Guerra GG, Joosten KF, Verbruggen SC, Van den Berghe G. Role of age of critically ill children at time of exposure to early or late parenteral nutrition in determining the impact hereof on long-term neurocognitive development: A secondary analysis of the PEPaNIC-RCT. Clin Nutr. 2021 Mar;40(3):1005-1012. doi: 10.1016/j.clnu.2020.07.004. Epub 2020 Jul 14. PMID 32758384
- [Derived] Jacobs A, Dulfer K, Eveleens RD, Hordijk J, Van Cleemput H, Verlinden I, Wouters PJ, Mebis L, Guerra GG, Joosten K, Verbruggen SC, Guiza F, Vanhorebeek I, Van den Berghe G. Long-term developmental effect of withholding parenteral nutrition in paediatric intensive care units: a 4-year follow-up of the PEPaNIC randomised controlled trial. Lancet Child Adolesc Health. 2020 Jul;4(7):503-514. doi: 10.1016/S2352-4642(20)30104-8. PMID 32562632
- [Derived] Hordijk J, Verbruggen S, Vanhorebeek I, Guiza F, Wouters P, Van den Berghe G, Joosten K, Dulfer K. Health-related quality of life of children and their parents 2 years after critical illness: pre-planned follow-up of the PEPaNIC international, randomized, controlled trial. Crit Care. 2020 Jun 16;24(1):347. doi: 10.1186/s13054-020-03059-2. PMID 32546247
- [Derived] van Puffelen E, Hulst JM, Vanhorebeek I, Dulfer K, Van den Berghe G, Joosten KFM, Verbruggen SCAT. Effect of late versus early initiation of parenteral nutrition on weight deterioration during PICU stay: Secondary analysis of the PEPaNIC randomised controlled trial. Clin Nutr. 2020 Jan;39(1):104-109. doi: 10.1016/j.clnu.2019.02.014. Epub 2019 Mar 4. PMID 30879734
- [Derived] van Puffelen E, Hulst JM, Vanhorebeek I, Dulfer K, Van den Berghe G, Verbruggen SCAT, Joosten KFM. Outcomes of Delaying Parenteral Nutrition for 1 Week vs Initiation Within 24 Hours Among Undernourished Children in Pediatric Intensive Care: A Subanalysis of the PEPaNIC Randomized Clinical Trial. JAMA Netw Open. 2018 Sep 7;1(5):e182668. doi: 10.1001/jamanetworkopen.2018.2668. PMID 30646158
- [Derived] Verstraete S, Verbruggen SC, Hordijk JA, Vanhorebeek I, Dulfer K, Guiza F, van Puffelen E, Jacobs A, Leys S, Durt A, Van Cleemput H, Eveleens RD, Garcia Guerra G, Wouters PJ, Joosten KF, Van den Berghe G. Long-term developmental effects of withholding parenteral nutrition for 1 week in the paediatric intensive care unit: a 2-year follow-up of the PEPaNIC international, randomised, controlled trial. Lancet Respir Med. 2019 Feb;7(2):141-153. doi: 10.1016/S2213-2600(18)30334-5. Epub 2018 Sep 14. PMID 30224325
- [Derived] Verstraete S, Vanhorebeek I, van Puffelen E, Derese I, Ingels C, Verbruggen SC, Wouters PJ, Joosten KF, Hanot J, Guerra GG, Vlasselaers D, Lin J, Van den Berghe G. Leukocyte telomere length in paediatric critical illness: effect of early parenteral nutrition. Crit Care. 2018 Feb 21;22(1):38. doi: 10.1186/s13054-018-1972-6. PMID 29463275
- [Derived] van Puffelen E, Polinder S, Vanhorebeek I, Wouters PJ, Bossche N, Peers G, Verstraete S, Joosten KFM, Van den Berghe G, Verbruggen SCAT, Mesotten D. Cost-effectiveness study of early versus late parenteral nutrition in critically ill children (PEPaNIC): preplanned secondary analysis of a multicentre randomised controlled trial. Crit Care. 2018 Jan 15;22(1):4. doi: 10.1186/s13054-017-1936-2. PMID 29335014
- [Derived] Fivez T, Kerklaan D, Mesotten D, Verbruggen S, Wouters PJ, Vanhorebeek I, Debaveye Y, Vlasselaers D, Desmet L, Casaer MP, Garcia Guerra G, Hanot J, Joffe A, Tibboel D, Joosten K, Van den Berghe G. Early versus Late Parenteral Nutrition in Critically Ill Children. N Engl J Med. 2016 Mar 24;374(12):1111-22. doi: 10.1056/NEJMoa1514762. Epub 2016 Mar 15. PMID 26975590
- [Derived] Fivez T, Kerklaan D, Verbruggen S, Vanhorebeek I, Verstraete S, Tibboel D, Guerra GG, Wouters PJ, Joffe A, Joosten K, Mesotten D, Van den Berghe G. Impact of withholding early parenteral nutrition completing enteral nutrition in pediatric critically ill patients (PEPaNIC trial): study protocol for a randomized controlled trial. Trials. 2015 May 1;16:202. doi: 10.1186/s13063-015-0728-8. PMID 25927936